CLINICAL TRIAL: NCT06842030
Title: Feasibility Trial of Darwin OncoTreat and OncoTarget Precision Medicine Testing to Improve Outcomes for Patients With Limited Metastatic Disease That Failed First-Line Systemic Therapy
Brief Title: Feasibility Trial of Darwin OncoTreat and OncoTarget Precision Medicine Testing
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Good Samaritan Hospital Medical Center, New York (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 24-002
Record Dates: First submitted 2025-01-07; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Personalized Medicine; Oligometastatic Disease; Feasibility

STUDY DESIGN:
Intervention Model Description: Feasibility of n=20
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Feasibility (Experimental): All study participants will get the same study intervention. It will include the usual radiation to all areas of visible disease. Systemic therapy will be determined by your medical oncologist with the supplemental information provided by the Darwin OncoTarget and OncoTreat test.
  Interventions: Diagnostic Test: Darwin OncoTarget and OncoTreat

INTERVENTIONS:
Diagnostic Test: Darwin OncoTarget and OncoTreat — Darwin OncoTarget and OncoTreat predict potential drugs with early markers of efficacy in early human clinical trials. Specifically, OncoTarget identifies high-affinity inhibitors of master regulator proteins, while OncoTreat identifies tumor-checkpoint module inhibitors that modulate the transcriptional activity of hyper-connected master regulators. These tests are now commercially available with Clinical Laboratory Improvement Amendments (CLIA) approval through Columbia Presbyterian Medical Center.

SUMMARY:
This is a feasibility trial to assess use of OncoTarget and OncoTreat testing in a basket design of patients with oligmetastasis across various solid tumor histology. Eligible oligometastatic patients that are receiving radiation therapy (n=20) will undergo mandatory tumor biopsy prior to precision medicine testing. Formalin fixed paraffin embedded tissue with >50% tumor will be sent to the Laboratory of Personalized Genomic Medicine at Columbia University Medical Center for Darwin OncoTarget and OncoTreat testing. This will be supplementing routine clinical care with the goal of improving outcomes. The treating oncologist will decide to administer standard of care systemic therapy or proceed with treatment recommended by precision medicine testing. Feasibility outcomes include the ability to have the OncoTarget and OncoTreat test performed based on tumor type and pathology, ability to procure agents, change in medication use, and identification of unknown barriers. This study is assessing the use of precision medicine in a population has documented poor outcomes with implications aimed at improving these outcomes.

DETAILED DESCRIPTION:
Despite significant progress in solid tumor oncology, including widespread genomic testing, metastatic cancer remains largely incurable and results in approximately 90% of cancer deaths. In the context of systems biology, RNA transcriptome-based (RNA-seq) testing is utilized to identify master regulator proteins that are putative drivers of tumor progression. After extensive preclinical testing and validation, Darwin OncoTarget and OncoTreat has been developed as a commercially available next generation precision oncology test with preliminary evidence of efficacy in treatment-refractory advanced cancers. We designed this pilot trial to assess the feasibility of integrating Darwin OncoTarget and OncoTreat testing in patients with oligometastases receiving comprehensive involved site radiotherapy.

Eligible patients are adults with solid tumor oligometastases with up to 10 discrete tumors amenable to radiation therapy following prior first-line systemic therapy. Tumor biopsy is required to allow for precision medicine testing to supplement standard clinical management. Formalin fixed paraffin embedded tissue with >50% tumor will be sent to the Laboratory of Personalized Genomic Medicine at Columbia University Medical Center for Darwin OncoTarget and OncoTreat testing. Patients will either continue standard of care systemic therapy or proceed with an alternative FDA approved treatment informed by Darwin testing. This trial evaluates the feasibility and utility of integrating novel precision oncology testing in a community hospital setting.

This study will utilize precision oncology testing in the population of induced, recurrent or persistent oligometastases that currently have limited or largely ineffective systemic treatment options. This trial represents an early attempt at integrating next generation precision medicine testing and systems biology in the context of radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients age ≥18 years with metastatic solid tumor who are candidates for comprehensive involved site radiotherapy to all areas of disease seen on whole body imaging.
* Patients with brain metastases are eligible provided they qualify as oligometastases (up to 10 lesions based on the SABR-COMET-10 trial) and are treatable with radiotherapy to all areas of visible disease.
* Patients with adequate bone marrow (absolute neutrophil ≥1000, hemoglobin ≥ 9 g/dl, platelets ≥100,000), kidney (creatinine ≤1.5 times upper limit of normal) and liver (bilirubin ≤1.5 times upper limit of normal).
* Patients being treated by radiation oncology at Good Samaritan University Hospital.

Exclusion Criteria:

* Patients with an estimated median survival of less than 6 months using the published and validated NEAT methodology.
* Patients who are pregnant and/or breast feeding or those with severe uncontrolled cardiac, pulmonary, infectious or organic brain disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-10 (Estimated); Primary Completion 2027-04-10 (Estimated); Study Completion 2027-04-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Test Performance Ability To Perform Test Versus Unable to Perform Test with Pathology Samples Needed >50% Tumor Tissue | Through study completion, an average of 2 years
  Proportion of participants whose tumor biopsy successfully undergoes OncoTarget and OncoTreat testing based on sufficient cellularity/DNA/RNA, defined as >50% tumor.
Feasibility: Percent Medication Change Versus No Medication Change Based on Treating Medical Oncologist Decision | Through study completion, an average of 2 years
  Percentage of participants whose chemotherapy management plan is changed based on the willingness of the medical oncologist to try at least one off-label medication recommended by Darwin testing.
Feasibility: Percent Medication Procured Through Insurance and/or Compassionate Use Versus Unable to Attain | Through study completion, an average of 2 years
  Out of the participants who are prescribed a drug from Darwin testing, the percentage that are procured FDA approved on-label and/or off-label agents through insurance or compassionate use in the setting of extensive preauthorization requirements prevalent in community oncology practice.
Feasibility: Qualitative Measurement of Barriers Noted Throughout Study | Through study completion, an average of 2 years
  Quantification and explanation of any unknown barriers that occur throughout the study process preventing an eligible participant from starting a drug recommended by Darwin testing.

SECONDARY OUTCOMES:
Systemic Therapy Change Compared to Standard of Care | Through study completion, an average of 2 years
  The proportion of cases where OncoTarget and OncoTreat testing, compared to standard of care genomic testing including Foundation One or Caris, results in a change in systemic treatment that can be implemented in a community hospital setting.
Progression-Free Survival | Patients will be followed as per standard of care, up to 5 years or until death. Event determined from date of enrollment until first documented progression or death from any cause, whichever came first, assessed up to 5 years.
  Progression-free survival defined as the time between enrollment and tumor progression or death for patients with oligometastases treated with comprehensive involved site radiotherapy compared to historical control patients treated without OncoTarget and OncoTreat testing.

CONTACTS AND LOCATIONS:
Locations (1):
- Good Samaritan University Hospital, West Islip, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pickert K: Is a Revolution in Cancer Treatment Within Reach? New York Times, 2023.
- [Background] Ganesh K, Massague J. Targeting metastatic cancer. Nat Med. 2021 Jan;27(1):34-44. doi: 10.1038/s41591-020-01195-4. Epub 2021 Jan 13. PMID 33442008
- [Background] Haslam A, Gill J, Prasad V. Estimation of the Percentage of US Patients With Cancer Who Are Eligible for Immune Checkpoint Inhibitor Drugs. JAMA Netw Open. 2020 Mar 2;3(3):e200423. doi: 10.1001/jamanetworkopen.2020.0423. PMID 32150268
- [Background] Haslam A, Kim MS, Prasad V. Updated estimates of eligibility for and response to genome-targeted oncology drugs among US cancer patients, 2006-2020. Ann Oncol. 2021 Jul;32(7):926-932. doi: 10.1016/j.annonc.2021.04.003. Epub 2021 Apr 20. PMID 33862157
- [Background] Kao J, Chen CT, Tong CC, Packer SH, Schwartz M, Chen SH, Sung MW. Concurrent sunitinib and stereotactic body radiotherapy for patients with oligometastases: final report of a prospective clinical trial. Target Oncol. 2014 Jun;9(2):145-53. doi: 10.1007/s11523-013-0280-y. Epub 2013 May 10. PMID 23660867
- [Background] Gomez DR, Tang C, Zhang J, Blumenschein GR Jr, Hernandez M, Lee JJ, Ye R, Palma DA, Louie AV, Camidge DR, Doebele RC, Skoulidis F, Gaspar LE, Welsh JW, Gibbons DL, Karam JA, Kavanagh BD, Tsao AS, Sepesi B, Swisher SG, Heymach JV. Local Consolidative Therapy Vs. Maintenance Therapy or Observation for Patients With Oligometastatic Non-Small-Cell Lung Cancer: Long-Term Results of a Multi-Institutional, Phase II, Randomized Study. J Clin Oncol. 2019 Jun 20;37(18):1558-1565. doi: 10.1200/JCO.19.00201. Epub 2019 May 8. PMID 31067138
- [Background] Palma DA, Olson R, Harrow S, Gaede S, Louie AV, Haasbeek C, Mulroy L, Lock M, Rodrigues GB, Yaremko BP, Schellenberg D, Ahmad B, Senthi S, Swaminath A, Kopek N, Liu M, Moore K, Currie S, Schlijper R, Bauman GS, Laba J, Qu XM, Warner A, Senan S. Stereotactic Ablative Radiotherapy for the Comprehensive Treatment of Oligometastatic Cancers: Long-Term Results of the SABR-COMET Phase II Randomized Trial. J Clin Oncol. 2020 Sep 1;38(25):2830-2838. doi: 10.1200/JCO.20.00818. Epub 2020 Jun 2. PMID 32484754
- [Background] Tsai CJ, Yang JT, Shaverdian N, Patel J, Shepherd AF, Eng J, Guttmann D, Yeh R, Gelblum DY, Namakydoust A, Preeshagul I, Modi S, Seidman A, Traina T, Drullinsky P, Flynn J, Zhang Z, Rimner A, Gillespie EF, Gomez DR, Lee NY, Berger M, Robson ME, Reis-Filho JS, Riaz N, Rudin CM, Powell SN; CURB Study Group. Standard-of-care systemic therapy with or without stereotactic body radiotherapy in patients with oligoprogressive breast cancer or non-small-cell lung cancer (Consolidative Use of Radiotherapy to Block [CURB] oligoprogression): an open-label, randomised, controlled, phase 2 study. Lancet. 2024 Jan 13;403(10422):171-182. doi: 10.1016/S0140-6736(23)01857-3. Epub 2023 Dec 14. PMID 38104577
- [Background] McBride S, Sherman E, Tsai CJ, Baxi S, Aghalar J, Eng J, Zhi WI, McFarland D, Michel LS, Young R, Lefkowitz R, Spielsinger D, Zhang Z, Flynn J, Dunn L, Ho A, Riaz N, Pfister D, Lee N. Randomized Phase II Trial of Nivolumab With Stereotactic Body Radiotherapy Versus Nivolumab Alone in Metastatic Head and Neck Squamous Cell Carcinoma. J Clin Oncol. 2021 Jan 1;39(1):30-37. doi: 10.1200/JCO.20.00290. Epub 2020 Aug 21. PMID 32822275
- [Background] Schoenfeld JD, Giobbie-Hurder A, Ranasinghe S, Kao KZ, Lako A, Tsuji J, Liu Y, Brennick RC, Gentzler RD, Lee C, Hubbard J, Arnold SM, Abbruzzese JL, Jabbour SK, Uboha NV, Stephans KL, Johnson JM, Park H, Villaruz LC, Sharon E, Streicher H, Ahmed MM, Lyon H, Cibuskis C, Lennon N, Jhaveri A, Yang L, Altreuter J, Gunasti L, Weirather JL, Mak RH, Awad MM, Rodig SJ, Chen HX, Wu CJ, Monjazeb AM, Hodi FS. Durvalumab plus tremelimumab alone or in combination with low-dose or hypofractionated radiotherapy in metastatic non-small-cell lung cancer refractory to previous PD(L)-1 therapy: an open-label, multicentre, randomised, phase 2 trial. Lancet Oncol. 2022 Feb;23(2):279-291. doi: 10.1016/S1470-2045(21)00658-6. Epub 2022 Jan 13. PMID 35033226
- [Background] Kao J, Sahagian M, Gupta V, Missios S, Sangal A. Long-term disease-free survival following comprehensive involved site radiotherapy for oligometastases. Front Oncol. 2023 Dec 5;13:1267626. doi: 10.3389/fonc.2023.1267626. eCollection 2023. PMID 38144534
- [Background] Antonia SJ, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Yokoi T, Chiappori A, Lee KH, de Wit M, Cho BC, Bourhaba M, Quantin X, Tokito T, Mekhail T, Planchard D, Kim YC, Karapetis CS, Hiret S, Ostoros G, Kubota K, Gray JE, Paz-Ares L, de Castro Carpeno J, Wadsworth C, Melillo G, Jiang H, Huang Y, Dennis PA, Ozguroglu M; PACIFIC Investigators. Durvalumab after Chemoradiotherapy in Stage III Non-Small-Cell Lung Cancer. N Engl J Med. 2017 Nov 16;377(20):1919-1929. doi: 10.1056/NEJMoa1709937. Epub 2017 Sep 8. PMID 28885881
- [Background] Kao J, Packer S, Vu HL, Schwartz ME, Sung MW, Stock RG, Lo YC, Huang D, Chen SH, Cesaretti JA. Phase 1 study of concurrent sunitinib and image-guided radiotherapy followed by maintenance sunitinib for patients with oligometastases: acute toxicity and preliminary response. Cancer. 2009 Aug 1;115(15):3571-80. doi: 10.1002/cncr.24412. PMID 19536893
- [Background] Tannock IF, Hickman JA. Limits to Personalized Cancer Medicine. N Engl J Med. 2016 Sep 29;375(13):1289-94. doi: 10.1056/NEJMsb1607705. No abstract available. PMID 27682039
- [Background] Le Tourneau C, Delord JP, Goncalves A, Gavoille C, Dubot C, Isambert N, Campone M, Tredan O, Massiani MA, Mauborgne C, Armanet S, Servant N, Bieche I, Bernard V, Gentien D, Jezequel P, Attignon V, Boyault S, Vincent-Salomon A, Servois V, Sablin MP, Kamal M, Paoletti X; SHIVA investigators. Molecularly targeted therapy based on tumour molecular profiling versus conventional therapy for advanced cancer (SHIVA): a multicentre, open-label, proof-of-concept, randomised, controlled phase 2 trial. Lancet Oncol. 2015 Oct;16(13):1324-34. doi: 10.1016/S1470-2045(15)00188-6. Epub 2015 Sep 3. PMID 26342236
- [Background] Chen AP, Kummar S, Moore N, Rubinstein LV, Zhao Y, Williams PM, Palmisano A, Sims D, O'Sullivan Coyne G, Rosenberger CL, Simpson M, Raghav KPS, Meric-Bernstam F, Leong S, Waqar S, Foster JC, Konate MM, Das B, Karlovich C, Lih CJ, Polley E, Simon R, Li MC, Piekarz R, Doroshow JH. Molecular Profiling-Based Assignment of Cancer Therapy (NCI-MPACT): A Randomized Multicenter Phase II Trial. JCO Precis Oncol. 2021 Jan 12;5:PO.20.00372. doi: 10.1200/PO.20.00372. eCollection 2021. PMID 33928209
- [Background] Prasad V. Perspective: The precision-oncology illusion. Nature. 2016 Sep 8;537(7619):S63. doi: 10.1038/537S63a. No abstract available. PMID 27602743
- [Background] Paull EO, Aytes A, Jones SJ, Subramaniam PS, Giorgi FM, Douglass EF, Tagore S, Chu B, Vasciaveo A, Zheng S, Verhaak R, Abate-Shen C, Alvarez MJ, Califano A. A modular master regulator landscape controls cancer transcriptional identity. Cell. 2021 Jan 21;184(2):334-351.e20. doi: 10.1016/j.cell.2020.11.045. Epub 2021 Jan 11. PMID 33434495
- [Background] Mundi PS, Dela Cruz FS, Grunn A, Diolaiti D, Mauguen A, Rainey AR, Guillan K, Siddiquee A, You D, Realubit R, Karan C, Ortiz MV, Douglass EF, Accordino M, Mistretta S, Brogan F, Bruce JN, Caescu CI, Carvajal RD, Crew KD, Decastro G, Heaney M, Henick BS, Hershman DL, Hou JY, Iwamoto FM, Jurcic JG, Kiran RP, Kluger MD, Kreisl T, Lamanna N, Lassman AB, Lim EA, Manji GA, McKhann GM, McKiernan JM, Neugut AI, Olive KP, Rosenblat T, Schwartz GK, Shu CA, Sisti MB, Tergas A, Vattakalam RM, Welch M, Wenske S, Wright JD, Canoll P, Hibshoosh H, Kalinsky K, Aburi M, Sims PA, Alvarez MJ, Kung AL, Califano A. A Transcriptome-Based Precision Oncology Platform for Patient-Therapy Alignment in a Diverse Set of Treatment-Resistant Malignancies. Cancer Discov. 2023 Jun 2;13(6):1386-1407. doi: 10.1158/2159-8290.CD-22-1020. PMID 37061969
- [Background] Guckenberger M, Lievens Y, Bouma AB, Collette L, Dekker A, deSouza NM, Dingemans AC, Fournier B, Hurkmans C, Lecouvet FE, Meattini I, Mendez Romero A, Ricardi U, Russell NS, Schanne DH, Scorsetti M, Tombal B, Verellen D, Verfaillie C, Ost P. Characterisation and classification of oligometastatic disease: a European Society for Radiotherapy and Oncology and European Organisation for Research and Treatment of Cancer consensus recommendation. Lancet Oncol. 2020 Jan;21(1):e18-e28. doi: 10.1016/S1470-2045(19)30718-1. PMID 31908301
- [Background] Kao J, Gold KD, Zarrili G, Copel E, Silverman AJ, Ramsaran SS, Yens D, Ryu S. Clinical Predictors of Survival for Patients with Stage IV Cancer Referred to Radiation Oncology. PLoS One. 2015 Apr 20;10(4):e0124329. doi: 10.1371/journal.pone.0124329. eCollection 2015. PMID 25894552
- [Background] Kao J, Eckardt P, Mceachron J, Atalla C, Sangal A. Predicting long-term survival following involved site radiotherapy for oligometastases. Oncol Lett. 2024 Jan 5;27(2):82. doi: 10.3892/ol.2024.14216. eCollection 2024 Feb. PMID 38249809
- [Background] Palma DA, Olson R, Harrow S, Correa RJM, Schneiders F, Haasbeek CJA, Rodrigues GB, Lock M, Yaremko BP, Bauman GS, Ahmad B, Schellenberg D, Liu M, Gaede S, Laba J, Mulroy L, Senthi S, Louie AV, Swaminath A, Chalmers A, Warner A, Slotman BJ, de Gruijl TD, Allan A, Senan S. Stereotactic ablative radiotherapy for the comprehensive treatment of 4-10 oligometastatic tumors (SABR-COMET-10): study protocol for a randomized phase III trial. BMC Cancer. 2019 Aug 19;19(1):816. doi: 10.1186/s12885-019-5977-6. PMID 31426760
- [Background] Zucker A, Tsai CJ, Loscalzo J, Calves P, Kao J. The NEAT Predictive Model for Survival in Patients with Advanced Cancer. Cancer Res Treat. 2018 Oct;50(4):1433-1443. doi: 10.4143/crt.2017.223. Epub 2018 Jan 24. PMID 29361815
- [Background] Casolino R, Beer PA, Chakravarty D, Davis MB, Malapelle U, Mazzarella L, Normanno N, Pauli C, Subbiah V, Turnbull C, Westphalen CB, Biankin AV. Interpreting and integrating genomic tests results in clinical cancer care: Overview and practical guidance. CA Cancer J Clin. 2024 May-Jun;74(3):264-285. doi: 10.3322/caac.21825. Epub 2024 Jan 4. PMID 38174605

DOCUMENTS (1):
  • Informed Consent Form (2024-03-13): https://cdn.clinicaltrials.gov/large-docs/30/NCT06842030/ICF_000.pdf